CLINICAL TRIAL: NCT01540227
Title: Penicillin Therapeutic Drug Monitoring in the Treatment of Infectious Syphilis. Do Low Serum Penicillin Levels Correlate With Treatment Failure?
Brief Title: Penicillin Therapeutic Drug Monitoring in the Treatment of Infectious Syphilis.
Status: Terminated | Type: Observational
Why Stopped: Low enrollment.
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: CIHR Canadian HIV Trials Network (Network)
Responsible Party: Principal Investigator, Paul MacPherson, Physician/Scientist, Ottawa Hospital Research Institute
Other Study IDs: CTN PT-011
Record Dates: First submitted 2012-02-16; First posted 2012-02-28 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Syphilis; Primary Syphilis; Secondary Syphilis; Early-Latent Syphilis
Keywords: Syphilis; Penicillin
MeSH Terms: conditions — Syphilis; Syphilis, primary; Syphilis, secondary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Syphilis Patients: Individuals presenting for treatment of primary, secondary or early latent syphilis at the Ottawa Hospital Immunodeficiency Clinic, the Ottawa Sexual Health Clinic or its satellite GayZone, the Montreal Chest Institute Immunodeficiency Clinic, or the Toronto General Immunodeficiency Clinic will be invited by their attending health care worker to participate in this study. Only patients presenting for and requiring treatment of infectious syphilis will be asked to participate.
  Interventions: Drug: Regular Treatment for Syphilis

INTERVENTIONS:
Drug: Regular Treatment for Syphilis — Drug: Benzathine Penicillin G (Bicillin)
  Dose: 2.4 million units
  Mode of Administration: intramuscular injection
  Duration of Treatment: one dose
  Health Canada approved indication: Yes

SUMMARY:
Syphilis is a sexually transmitted infection that causes genital sores and rash, but in some circumstances may result in more severe and unexpected symptoms. These severe symptoms could include eye infections, meningitis (infection of the membranes covering the brain and spinal cord), and liver infection. If not properly treated, syphilis can also lead to heart problems and dementia (a decline in reasoning, memory and other mental abilities) years down the road. There has been an increase in the number of reported cases of syphilis in North America, Europe, and Australia over the past decade. The number of new syphilis infections in Canada has increased roughly 10-fold over the past 10 years.

Since 1943, the antibiotic penicillin has been used to treat syphilis; however, very little information has been gathered to determine the proper dose of penicillin or appropriate duration of treatment. Added to this, several studies have shown that the recommended dose of penicillin fails to cure syphilis in 20-30% of patients. Since the number of people infected with syphilis is increasing, and since syphilis has the potential to cause serious disease, the investigators need better information on how to treat syphilis effectively.

This study aims to determine whether the current dose of penicillin recommended to treat syphilis is sufficient to cure the infection. Specifically the investigators will try to determine whether the amount of penicillin in your blood 3 and 7 days after receiving treatment for syphilis is sufficient to cure the infection as demonstrated by a blood test 6 or 12 months from now. This study is a multi-centered trial based in Ottawa but with centers recruiting both in Montreal and Toronto. A total of 120 participants with syphilis will be recruited into this study. The treatment you will receive for syphilis in this study does not differ from that you would receive normally; the investigators are only observing the levels of penicillin in your blood and relating them with the outcome of treatment.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be considered eligible for entry into the study:

1. At least 18 years of age
2. Presenting with clinical signs of either primary or secondary syphilis; or with early latent syphilis and documented negative serology within the past 12 months.
3. Positive syphilis serology (reactive CMIA and TP-PA) with a defined RPR titer at the time of diagnosis and enrolment
4. Able to provide informed consent
5. Able to communicate in either English of French
6. Able to return for follow-up

Exclusion Criteria:

Participants are not eligible to participate in the study if any of the following conditions are met:

1. Diagnosis of late latent syphilis, tertiary syphilis, or syphilis of unknown duration
2. Allergy to penicillin
3. Diagnosis of neurosyphilis requiring treatment with intravenous penicillin
4. Treatment with doxycycline or ceftriaxone
5. Treatment with more than one intramuscular dose of benzathine penicillin G
6. Treatment with any antibiotics within the 6 weeks prior to enrolment
7. Pregnant or breastfeeding
8. Any immune modulating therapy
9. Patient is unable or unwilling to return for blood sampling at 3 and 7 days post treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals presenting for treatment of primary, secondary or early latent syphilis will be invited by their attending health care worker to participate in this study. Only patients presenting for and requiring treatment of infectious syphilis will be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2016-11-10 (Actual); Study Completion 2016-11-10 (Actual)

PRIMARY OUTCOMES:
Penicillin and Treatment Failure | 6 months post-treatment
  To determine if serum penicillin concentrations measured at days 3 and 7 post-treatment differ between those who achieve successful treatment of infectious syphilis versus those who experience treatment failure.

SECONDARY OUTCOMES:
HIV and Treatment Failure | 6 months post-treatment
  To determine if serum penicillin levels and treatment failures differ between HIV-positive and HIV-negative individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Paul A MacPherson, MD/PhD, Principal Investigator — The Ottawa Hospital/The University of Ottawa/OHRI
Locations (3):
- Canada (3):
  - The Ottawa Hospital, Ottawa, Ontario
  - Ottawa Sexual Health Clinic/GayZone, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario